CLINICAL TRIAL: NCT04642365
Title: An Open-Label, Multicenter, Phase Ib Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Anti-Tumor Activity of RO7296682 in Combination With Atezolizumab in Participants With Advanced and/or Metastatic Solid Tumors
Brief Title: A Study to Evaluate the Safety and Tolerability of RO7296682 in Combination With Atezolizumab in Participants With Advanced Solid Tumors.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor decided to terminate the study early, due to recruitment challenges for Part II and, based on the totality of data generated with a low likelihood of achieving the targeted efficacy, to open Part III.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP42595; 2020-003164-82 (EudraCT Number)
Record Dates: First submitted 2020-11-23; First posted 2020-11-24 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumors
Keywords: RG6292
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part I (Experimental): Dose-Escalation: Mixed solid tumors participants will receive ascending doses of RO7296682 with a fixed dose of Atezolizumab, every three weeks (Q3W) until either the Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D) is defined.
  Interventions: Drug: RO7296682; Drug: Atezolizumab
- Part II (Experimental): Dose-Expansion: Will start once MTD/RP2D dose of RO7296682 in combination with Atezolizumab is defined in Part I. Participants with selected tumor types will receive a fixed dose of RO7296682 in combination with Atezolizumab.
  Interventions: Drug: RO7296682; Drug: Atezolizumab
- Part III (Exploratory) (Experimental): Dose-Expansion: Will start once MTD/RP2D dose of RO7296682 in combination with Atezolizumab is defined in Part I and if clinical activity is seen in this trial or in the single agent study (WP41188). Participants with selected tumor types will receive a fixed dose of RO7296682 in combination with Atezolizumab at the dosing regimen established in Part I.
  Interventions: Drug: RO7296682; Drug: Atezolizumab

INTERVENTIONS:
Drug: RO7296682 — RO7296682 will be administered as per the schedules specified in the respective arms.
Drug: Atezolizumab — Atezolizumab will be administered as per the schedules specified in the respective arms.

SUMMARY:
This study will evaluate the safety, tolerability and preliminary anti-tumor activity of RO7296682 in combination with Atezolizumab in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of advanced and/or metastatic solid tumors who have progressed on a standard therapy, are intolerant to standard of care (SoC), and/or and non-amenable to SoC.

Participants whose tumors have known sensitizing mutations must have experienced disease progression (during or after treatment) or intolerance to treatment with a respective targeted therapy.

* Measurable disease according to RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Able to provide the most recent archival tumor tissue samples.
* Adequate cardiovascular, haematological, liver and renal function.
* Participants on therapeutic anticoagulation must be on a stable anticoagulant regimen.
* Women of Childbearing Potential: Agreement to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive methods.
* Men: Agreement to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive methods and refrain from donating sperm.

Exclusion Criteria:

* Pregnancy, lactation, or breastfeeding.
* Known hypersensitivity to any of the components of RO7296682 and atezolizumab, including but not limited to hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies.
* History or clinical evidence of central nervous system (CNS) primary tumors or metastases.
* Participants with another invasive malignancy in the last two years.
* Participants with known active or uncontrolled infection.
* Positive HIV test at screening.
* Positive for Hepatitis B and C.
* Vaccination with live vaccines within 28 days prior to C1D1.
* Major surgical procedure or significant traumatic injury within 28 days prior to first RO7296682 and atezolizumab infusion.
* Participants with wound healing complications.
* Dementia or altered mental status that would prohibit informed consent.
* History of Stevens-Johnson syndrome, toxic epidermal necrolysis, or DRESS (drug rash with eosinophilia and systemic symptoms).
* Active or history of autoimmune disease or immune deficiency.
* Prior treatment with CPIs (e.g. anti-CTLA4, anti-PD1, anti-PDL1), immunomodulatory monoclonal antibodies (mAbs) and/or mAb-derived therapies (approved or investigational) is approved.
* Treatment with standard radiotherapy, any chemotherapeutic agent, targeted therapy or treatment with any other investigational drug (defined as treatment for which there is currently no regulatory authority-approved indication) within 28 days or 5 half-lives of the drug (whichever is shorter), prior to the first RO7296882 administration on C1D1.
* Radiotherapy within the last 4 weeks before start of study drug treatment, with the exception of limited palliative radiotherapy (for which no wash out period is required).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- MD Anderson Cancer Center, Houston, Texas, United States
- Peter Maccallum Cancer Institute, Melbourne, Victoria, Australia
- Cliniques Universitaires St-Luc, Brussels, Belgium
- Canada (3):
  - BC Cancer Agency - Vancouver, Vancouver, British Columbia
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Rigshospitalet, København Ø, Denmark
- Spain (3):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 49 participants took part in the study across 10 investigative sites in 6 countries. This study was planned to be conducted in 3 parts. Part 1 (Dose-escalation): ascending doses of RO7296682 + fixed dose of atezolizumab, Part 2 (Dose expansion): fixed dose of RO7296682 + atezolizumab and Part 3 (Exploratory). Part 2 was prematurely terminated and Part 3 was not opened for enrollment due to study termination.
Pre-assignment Details: Participants with advanced and/or metastatic non-small cell lung cancer (NSCLC), melanoma (MEL), head and neck squamous cell carcinoma (HNSCC), esophageal cancer (EsC), triple-negative breast cancer (TNBC), and ovarian cancer (OvCa) who progressed on all standard therapies, were intolerant to standard of care (SoC), and/or were non-amenable to SoC/for whom SoC did not exist were enrolled in Part 1 cohorts.
Groups:
- Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg: Participants received RO7296682, 0.3 milligrams (mg) as an intravenous (IV) infusion in combination with atezolizumab, 1200 mg, as an IV infusion every 3 week (Q3W) for a maximum of 13.2 months.
- Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg: Participants received RO7296682, 1.5 mg, as an IV infusion in combination with atezolizumab, 1200 mg, as an IV infusion Q3W for a maximum of 23.7 months.
- Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg: Participants received RO7296682, 9 mg, as an IV infusion in combination with atezolizumab, 1200 mg, as an IV infusion Q3W for a maximum of 12 months.
- Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg: Participants received RO7296682, 20 mg, as an IV infusion in combination with atezolizumab, 1200 mg, as an IV infusion Q3W for a maximum of 16.6 months.
- Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg: Participants received RO7296682, 40 mg, as an IV infusion in combination with atezolizumab, 1200 mg, as an IV infusion Q3W for a maximum of 8.6 months.
- Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg: Participants received RO7296682, 80 mg, as an IV infusion in combination with atezolizumab, 1200 mg, as an IV infusion Q3W for a maximum of 24 months.
- Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg: Participants received RO7296682, 160 mg, as an IV infusion in combination with atezolizumab, 1200 mg, as an IV infusion Q3W for a maximum of 2.8 months.
- Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg: Participants with advanced and/or metastatic NSCLC, MEL, HNSCC with inflamed tumor phenotype and acquired resistance to most recent programmed death protein 1 (PD-1) or programmed death ligand 1 (PD-L1) treatment received RO7296682, 70 mg, as an IV infusion in combination with atezolizumab, 1200 mg, as an IV infusion Q3W for a maximum of 5.5 months.
Period: Overall Study
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg
Started | 6 | 6 | 7 | 7 | 7 | 6 | 7 | 3
Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not Completed | 6 | 6 | 7 | 7 | 6 | 6 | 7 | 3
Not completed — Death | 3 | 2 | 4 | 5 | 5 | 3 | 2 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Study Terminated By Sponsor | 0 | 2 | 1 | 1 | 1 | 2 | 2 | 1
Not completed — Symptomatic Deterioration | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study treatment, whether prematurely withdrawn from the study or not.
Groups:
- Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg: Participants received RO7296682, 0.3 mg as an IV infusion in combination with atezolizumab, 1200 mg, as an IV infusion Q3W for a maximum of 13.2 months.
- Total: Total of all reporting groups
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg | Total
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 7 | 6 | 7 | 3 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (12.4) | 61.7 (10.5) | 62.6 (10.1) | 62.0 (13.3) | 66.4 (9.7) | 63.0 (10.9) | 57.1 (9.7) | 55.3 (8.6) | 60.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 4 | 3 | 2 | 5 | 1 | 23
  Male | 3 | 4 | 4 | 3 | 4 | 4 | 2 | 2 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 6 | 6 | 7 | 6 | 6 | 5 | 7 | 3 | 46
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 6 | 7 | 6 | 6 | 6 | 7 | 3 | 47
  Missing | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and regardless of a causal relationship with this treatment. An AE can therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with use of investigational product, whether or not considered related to investigational product.
Time Frame: From Day 1 up to the end of safety follow-up (up to 28.5 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 7 | 6 | 7
Participants | 6 | 6 | 7 | 7 | 7 | 5 | 7

2. Primary Outcome: Part 2: Number of Participants With AEs
Description: as for outcome 1
Time Frame: From Day 1 up to the end of safety follow-up (up to 9.3 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 3
Participants | 3

3. Primary Outcome: Part 1: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as the occurrence of any of the following toxicities related to RO7296682 and atezolizumab that occurs during the DLT assessment window and not attributable to the underlying disease or an intercurrent illness: Any Grade ≥ 3 hematologic toxicity; Any Grade ≥ 3 non-hematologic toxicity; any other RO7296682-related toxicity considered significant enough to qualify as a DLT in the opinion of the Investigator and after discussion with the Sponsor.
Time Frame: From Cycle 1 Day 1 up Cycle 2 Day 8 (1 Cycle = 21 days)
Population: DLT evaluable population included participants who completed the DLT period with two administrations of RO7296682/atezolizumab without DLT, or participants reported with a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 7 | 6 | 7
Participants | 0 | 0 | 0 | 1 | 0 | 1 | 0

4. Primary Outcome: Part 2: Objective Response Rate (ORR)
Description: ORR was determined as the percentage of participants with an overall response (OR) of complete response (CR) or partial response (PR) as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters (SOD) of target lesions, taking as reference the baseline SOD. Percentages have been rounded off to the nearest decimal point.
Time Frame: Part 2: From Day 1 up to end of safety follow-up (up to 9.3 months)
Population: Efficacy population included all participants who received at least one dose of RO7296682 in combination with atezolizumab, and who had at least one baseline and one on-study tumor assessment and discontinued the study because of progression before the first on-study tumor assessment were considered response evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 3
percentage of participants | 0 [0 to 70.76]

5. Secondary Outcome: Part 1: ORR
Description: ORR was determined as the percentage of participants with an OR of CR or PR as determined by the investigator using RECIST v.1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. Percentages have been rounded off to the nearest decimal point.
Time Frame: From Day 1 up to end of safety follow-up (up to 28.5 months)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 5 | 6 | 7 | 7 | 7 | 6 | 7
percentage of participants | 0 [0 to 52.18] | 0 [0 to 45.93] | 0 [0 to 40.96] | 0 [0 to 40.96] | 28.6 [3.67 to 70.96] | 16.7 [0.42 to 64.12] | 0 [0 to 40.96]

6. Secondary Outcome: Part 1 and 2: Disease Control Rate (DCR)
Description: DCR was determined as the rate of participants with an OR of either CR, PR, or stable disease (SD) rate as determined by the investigator using RECIST v.1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD). PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on the study including baseline (nadir). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Percentages have been rounded off to the nearest decimal point.
Time Frame: Part 1: From Day 1 up to end of safety follow-up (up to 28.5 months); Part 2: From Day 1 up to end of safety follow-up (up to 9.3 months)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 5 | 6 | 7 | 7 | 7 | 6 | 7 | 3
percentage of participants | 40.0 [5.27 to 85.34] | 33.3 [4.33 to 77.72] | 57.1 [18.41 to 90.10] | 42.9 [9.90 to 81.59] | 71.4 [29.04 to 96.33] | 66.7 [22.28 to 95.67] | 14.3 [0.36 to 57.87] | 33.3 [0.84 to 90.57]

7. Secondary Outcome: Part 1 and 2: Duration of Response (DoR)
Description: DOR was calculated for participants who had a best OR of CR/PR. DOR was defined as time from first occurrence of a documented OR until the time of documented PD or death from any cause, whichever occurs first. CR=the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR=at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. PD=at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on the study including baseline (nadir). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Participants without PD/death (within 30 days from last treatment) were censored on the last day of tumor assessment. Participants without post-baseline (PB) or with all PB assessments but known to be alive were censored at the date of study treatment initiation plus one day.
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
days |  |  |  |  | 156 [105.0 to 207.0] | 364.00 [364.0 to 364.0] |  |

8. Secondary Outcome: Part 1 and 2: Progression-Free Survival (PFS)
Description: PFS was defined as the time from study treatment initiation to the first occurrence of documented PD (per RECIST v1.1) or death from any cause, whichever occurs first. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on the study including baseline (nadir). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Participants without PD or death (within 30 days from last treatment) were censored at the last day of tumor assessment. Participants without PB or with all PB assessments but known to be alive were censored at the date of study treatment initiation plus one day.
Time Frame: as for outcome 6
Population: Efficacy population included all participants who received at least one dose of RO7296682 in combination with atezolizumab, and who had at least one baseline and one on-study tumor assessment and discontinued the study because of progression before the first on-study tumor assessment were considered response evaluable. Overall number analyzed is the number of participants with data available for analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 5 | 6 | 6 | 7 | 7 | 4 | 6 | 3
days | 52.0 [23.0 to NA] — The upper limit of the 95% confidence interval (CI) was not estimable due to insufficient number of participants with events. | 58.0 [56.0 to 103.0] | 121.0 [70.0 to 148.0] | 59.0 [31.0 to 225.0] | 135.0 [53.0 to 182.0] | 111.0 [105.0 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events. | 51.5 [46.0 to 57.0] | 69.0 [57.0 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events.

9. Secondary Outcome: Part 1 and 2: Overall Survival (OS)
Description: OS was defined as the time from the first dose of study treatment to the time of death from any cause. Participants who were still alive at the time of analysis were censored at the time of their last study assessment (for active participants) or at the last date known alive (for participants in follow-up).
Time Frame: Part 1: From Day 1 up to end of survival follow-up (36 months); Part 2: From Day 1 up to end of safety follow-up (up to 9.3 months)
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 5 | 4 | 4 | 5 | 5 | 3 | 3 | 2
days | 181.0 [36.0 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events. | 295.0 [84.0 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events. | 352.0 [263.0 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events. | 237.0 [213.0 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events. | 353.0 [129.0 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events. | 230.0 [111.0 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events. | 304.0 [137.0 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events. | 73.0 [69.0 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events.

10. Secondary Outcome: Part 1 and 2: Area Under the Curve From Time of Dosing to the Last Timepoint at the End of the Dosing Period (AUClast) of RO7296682
Time Frame: Cycles 1 and 4: Predose, end of infusion, and at 24, 72, 168, and 336 hours post-dose (1 Cycle = 21 days)
Population: PK-evaluable population included all participants who received at least one dose of study treatment and who had data from at least one post-dose sample. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*micrograms/milliliters (h*μg/mL)
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 7 | 6 | 7 | 3
hours*micrograms/milliliters (h*μg/mL)
  Cycle 1 | 14.3 (89.3) | 83.7 (50.2) | 507 (43.9) | 1050 (26.9) | 2100 (50.8) | 3860 (22.3) | 9890 (23.8) | NA (NA) — Samples were below the limit of quantification, hence geometric mean and geometric coefficient of variation were unevaluable.
  Cycle 4: number analyzed (Participants) | 4 | 3 | 5 | 2 | 5 | 2 | 2 | 3
  Cycle 4 | 19.4 (79.8) | 109 (34.9) | 599 (45.3) | 1130 (146) | 2780 (82.5) | 5460 (8.20) | 16700 (0.708) | NA (NA) — Samples were below the limit of quantification, hence geometric mean and geometric coefficient of variation were unevaluable.

11. Secondary Outcome: Part 1 and 2: Maximum Concentration (Cmax) of RO7296682
Time Frame: Cycles 1 and 4: Predose, end of infusion, and at 24, 72, 168, and 336 hours post-dose (1 Cycle = 21 days)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliters (μg/mL)
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 7 | 6 | 7 | 3
micrograms/milliliters (μg/mL)
  Cycle 1 | 0.0921 (54.1) | 0.555 (22.2) | 3.18 (19.3) | 8.23 (32.8) | 12.7 (40.9) | 27.3 (34.5) | 61.7 (17.5) | NA (NA) — Samples were below the limit of quantification, hence geometric mean and geometric coefficient of variation were unevaluable.
  Cycle 4: number analyzed (Participants) | 4 | 3 | 5 | 2 | 5 | 2 | 2 | 3
  Cycle 4 | 0.119 (66.3) | 0.544 (28.8) | 3.27 (21.0) | 7.82 (40.4) | 15.3 (43.9) | 34.2 (27.8) | 85.2 (4.32) | NA (NA) — Samples were below the limit of quantification, hence geometric mean and geometric coefficient of variation were unevaluable.

12. Secondary Outcome: Part 1 and 2: Time of Maximum Concentration (Tmax) of RO7296682
Time Frame: Cycles 1 and 4: Predose, end of infusion, and at 24, 72, 168, and 336 hours post-dose (1 Cycle = 21 days)
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 7 | 6 | 7 | 3
hours
  Cycle 1 | 5.53 [4.12 to 6.75] | 4.15 [4.00 to 7.28] | 4.17 [3.92 to 19.9] | 4.92 [4.00 to 6.67] | 4.07 [4.00 to 7.00] | 4.07 [4.00 to 26.0] | 4.13 [4.00 to 5.67] | NA [NA to NA] — Samples were below the limit of quantification, hence median and full range were unevaluable.
  Cycle 4: number analyzed (Participants) | 4 | 3 | 5 | 2 | 5 | 2 | 2 | 3
  Cycle 4 | 1.41 [1.00 to 4.00] | 1.17 [1.00 to 4.08] | 1.15 [1.05 to 2.93] | NA [1.05 to 23.0] — Median values cannot be derived for two participants. | 1.17 [1.00 to 3.75] | NA [1.22 to 3.50] — Median values cannot be derived for two participants. | NA [1.08 to 1.27] — Median values cannot be derived for two participants. | NA [NA to NA] — Samples were below the limit of quantification, hence median and full range were unevaluable.

13. Secondary Outcome: Part 1 and 2: Volume of Distribution at Steady State Conditions (Vss) of RO7296682
Time Frame: Cycles 1 and 4: Predose, end of infusion, and at 24, 72, 168, and 336 hours post-dose (1 Cycle = 21 days)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre (L)
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 7 | 6 | 7 | 3
Litre (L)
  Cycle 1 | 6.91 (49.8) | 5.41 (16.9) | 5.31 (33.6) | 5.94 (12.8) | 7.29 (45.3) | 6.14 (50.7) | 5.84 (42.1) | NA (NA) — Samples were below the limit of quantification, hence geometric mean and geometric coefficient of variation were unevaluable.
  Cycle 4: number analyzed (Participants) | 4 | 3 | 5 | 2 | 5 | 2 | 2 | 3
  Cycle 4 | 5.75 (142) | 6.12 (19.4) | 5.59 (41.3) | 6.50 (10.5) | 5.59 (44.8) | 3.96 (24.2) | 5.22 (5.82) | NA (NA) — Samples were below the limit of quantification, hence geometric mean and geometric coefficient of variation were unevaluable.

14. Secondary Outcome: Part 1 and 2: Half-life (t~1/2) of RO7296682
Time Frame: Cycles 1 and 4: Predose, end of infusion, and at 24, 72, 168, and 336 hours post-dose (1 Cycle = 21 days)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 7 | 6 | 7 | 3
days
  Cycle 1 | 10.1 (40.2) | 8.89 (32.8) | 8.91 (29.7) | 9.43 (31.1) | 10.8 (21.6) | 9.15 (42.4) | 11.2 (49.7) | NA (NA) — Samples were below the limit of quantification, hence geometric mean and geometric coefficient of variation were unevaluable.
  Cycle 4: number analyzed (Participants) | 4 | 3 | 5 | 2 | 5 | 2 | 2 | 3
  Cycle 4 | 10.3 (25.3) | 13.2 (53.0) | 10.8 (51.2) | 12.1 (109) | 9.65 (32.1) | 7.92 (3.64) | 15.3 (4.28) | NA (NA) — Samples were below the limit of quantification, hence geometric mean and geometric coefficient of variation were unevaluable.

15. Secondary Outcome: Part 1: Serum Concentration of Atezolizumab
Description: 1 Cycle = 21 days.
Time Frame: Predose on Day 1 of Cycles 1 to 9, 12, 14, and 17; End of infusion (EOI) on Day 1 of Cycles 1 and 4; end of study/early discontinuation (up to 28.5 months)
Population: PK-evaluable population included all participants who received at least one dose of study treatment and who had data from at least one post-dose sample. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 7 | 6 | 5 | 2
μg/mL
  Cycle 1 Day 1 Predose | NA (NA) — Geometric Mean and Geometric Coefficient of Variation was not estimable as samples were below limit of quantification (BLQ). | NA (NA) — Geometric Mean and Geometric Coefficient of Variation was not estimable as samples were BLQ. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation was not estimable as samples were BLQ. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation was not estimable as samples were BLQ. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation was not estimable as samples were BLQ. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation was not estimable as samples were BLQ. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation was not estimable as samples were BLQ. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation was not estimable as samples were BLQ.
  Cycle 1 Day 1 - EOI: number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 6 | 5 | 2
  Cycle 1 Day 1 - EOI | 432 (25.9) | 387 (17.7) | 427 (32.4) | 374 (19.5) | 363 (29.5) | 379 (23.3) | 492 (13.1) | 410 (25.8)
  Cycle 2 Day 1 - Predose: number analyzed (Participants) | 6 | 6 | 6 | 3 | 7 | 4 | 5 | 0
  Cycle 2 Day 1 - Predose | 65.7 (91.5) | 74.6 (44.6) | 98.2 (39.4) | 65.8 (21.6) | 58.0 (72.2) | 67.4 (50.0) | 87.9 (46.3) |
  Cycle 3 Day 1 Predose: number analyzed (Participants) | 4 | 5 | 4 | 3 | 7 | 2 | 2 | 0
  Cycle 3 Day 1 Predose | 153 (32.4) | 177 (75.2) | 89.9 (98.8) | 84.0 (49.1) | 121 (35.5) | 82.4 (39.8) | 181 (35.1) |
  Cycle 4 Day 1 Predose: number analyzed (Participants) | 4 | 3 | 4 | 1 | 5 | 3 | 2 | 0
  Cycle 4 Day 1 Predose | 180 (29.2) | 131 (29.1) | 130 (41.7) | NA (NA) — Since only 1 participant was evaluable, Geometric mean (GM) and Geometric Coefficient of Variation could not be estimated. | 159 (42.5) | 115 (56.4) | 260 (16.9) |
  Cycle 4 Day 1 - EOI Atezo: number analyzed (Participants) | 3 | 3 | 3 | 1 | 5 | 3 | 1 | 0
  Cycle 4 Day 1 - EOI Atezo | 566 (15.7) | 527 (8.40) | 450 (28.0) | NA (NA) — Since only 1 participant was evaluable, GM and Geometric Coefficient of Variation could not be estimated. | 512 (35.9) | 510 (14.8) | NA (NA) — Since only 1 participant was evaluable, GM and Geometric Coefficient of Variation could not be estimated. |
  Cycle 5 Day 1 Predose: number analyzed (Participants) | 4 | 3 | 4 | 1 | 4 | 2 | 0 | 0
  Cycle 5 Day 1 Predose | 194 (40.9) | 153 (33.0) | 151 (60.0) | NA (NA) — Since only 1 participant was evaluable, GM and Geometric Coefficient of Variation could not be estimated. | 190 (31.6) | 162 (26.4) |  |
  Cycle 6 Day 1 Predose: number analyzed (Participants) | 2 | 2 | 4 | 1 | 3 | 2 | 0 | 0
  Cycle 6 Day 1 Predose | 194 (11.7) | 139 (112) | 160 (51.1) | NA (NA) — Since only 1 participant was evaluable, GM and Geometric Coefficient of Variation could not be estimated. | 237 (23.4) | 169 (44.8) |  |
  Cycle 7 Day 1 Predose: number analyzed (Participants) | 1 | 2 | 3 | 0 | 2 | 1 | 0 | 0
  Cycle 7 Day 1 Predose | NA (NA) — Since only 1 participant was evaluable, GM and Geometric Coefficient of Variation could not be estimated. | 201 (52.4) | 154 (64.5) |  | 265 (9.61) | NA (NA) — Since only 1 participant was evaluable, GM and Geometric Coefficient of Variation could not be estimated. |  |
  Cycle 8 Day 1 Predose: number analyzed (Participants) | 1 | 2 | 1 | 0 | 2 | 0 | 0 | 0
  Cycle 8 Day 1 Predose | NA (NA) — Since only 1 participant was evaluable, GM and Geometric Coefficient of Variation could not be estimated. | 209 (36.0) | NA (NA) — Since only 1 participant was evaluable, GM and Geometric Coefficient of Variation could not be estimated. |  | 238 (39.0) |  |  |
  Cycle 9 Day 1 Predose: number analyzed (Participants) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
  Cycle 9 Day 1 Predose | NA (NA) — Since only 1 participant was evaluable, GM and Geometric Coefficient of Variation could not be estimated. | NA (NA) — Since only 1 participant was evaluable, GM and Geometric Coefficient of Variation could not be estimated. | NA (NA) — Since only 1 participant was evaluable, GM and Geometric Coefficient of Variation could not be estimated. |  | NA (NA) — Since only 1 participant was evaluable, GM and Geometric Coefficient of Variation could not be estimated. |  |  |
  Cycle 12 Day 1 Predose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 12 Day 1 Predose | NA (NA) — Since only 1 participant was evaluable, GM and Geometric Coefficient of Variation could not be estimated. |  |  |  |  |  |  |
  Cycle 14 Day 1 Predose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 14 Day 1 Predose | NA (NA) — Since only 1 participant was evaluable, GM and Geometric Coefficient of Variation could not be estimated. |  |  |  |  |  |  |
  Cycle 17 Day 1 Predose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 17 Day 1 Predose | NA (NA) — Since only 1 participant was evaluable, GM and Geometric Coefficient of Variation could not be estimated. |  |  |  |  |  |  |
  End of Study: number analyzed (Participants) | 3 | 2 | 5 | 3 | 3 | 1 | 2 | 0
  End of Study | 135 (37.9) | 105 (37.4) | 141 (34.0) | 74.1 (21.1) | 112 (16.4) | NA (NA) — Since only 1 participant was evaluable, GM and Geometric Coefficient of Variation could not be estimated. | 61.3 (13.0) |

16. Secondary Outcome: Part 1 and 2: Number of Participants With Treatment-induced Changes in T Regulatory C Ells (Treg) Levels in Blood and/or Tumor as Compared to Baseline
Description: Treg depletion was defined as a reduction to 25% of baseline. As pre-specified in the protocol, the sponsor had the discretion to discontinue any part of the study at any time. On October 3, 2022, the sponsor decided to terminate Part 2 early due to recruitment challenges. As only 3 participants were enrolled in Part 2: Cohort 1, the sponsor decided not to collect and analyze data for the pharmacodynamic endpoints in Part 2.
Time Frame: Baseline up to 28 days post last dose (up to 24.9 months)
Population: Pharmacodynamic (PD) evaluable population included all participants who had at least one pre-dose and one post-dose PD assessment were included and analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 7 | 6 | 7 | 0
Participants | 1 | 1 | 5 | 5 | 7 | 5 | 3 |

17. Secondary Outcome: Part 1 and 2: Treatment-induced Changes in Teff (T-effector Cell)/Treg Ratio in Blood and/or Tumor as Compared to Baseline
Description: As pre-specified in the protocol, the sponsor had the discretion to discontinue any part of the study at any time. On October 3, 2022, the sponsor decided to terminate Part 2 early due to recruitment challenges. As only 3 participants were enrolled in Part 2: Cohort 1, the sponsor decided not to collect and analyze data for the pharmacodynamic endpoints in Part 2.
Time Frame: Cycle 1 Day 1 (end of infusion [EOI]); Cycle 1 Day 4 (72 hours post dose); Cycle 1 Day 8 (168 hours post dose); Cycle 1 Day 15 (336 hours post dose)
Population: Pharmacodynamic (PD) evaluable population included all participants who had at least one pre-dose and one post-dose PD assessment were included and analyzed according to the treatment they actually received. Number analyzed per timepoint are unique number of participants out all the assessed participants with data available for analysis at the specified timepoint. Different participants may have contributed data for each timepoint.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 7 | 6 | 7 | 0
ratio
  Cycle 1 Day 1 (EOI): number analyzed (Participants) | 5 | 3 | 5 | 5 | 6 | 6 | 2 | 0
  Cycle 1 Day 1 (EOI) | 1.59 (1.43) | 0.83 (0.67) | 0.41 (0.15) | 0.27 (0.20) | 0.37 (0.60) | 0.68 (0.92) | 0.32 (0.12) |
  Cycle 1 Day 4 (72 hours Post-dose): number analyzed (Participants) | 5 | 1 | 5 | 6 | 4 | 6 | 2 | 0
  Cycle 1 Day 4 (72 hours Post-dose) | 0.69 (0.78) | 0.17 (NA) — Since only 1 participant was evaluated, standard deviation could not be calculated. | 0.30 (0.12) | 0.60 (1.06) | 0.19 (0.22) | 0.29 (0.31) | 0.52 (0.47) |
  Cycle 1 Day 8 (168 hours Post-dose): number analyzed (Participants) | 2 | 2 | 5 | 6 | 5 | 5 | 3 | 0
  Cycle 1 Day 8 (168 hours Post-dose) | 1.55 (1.37) | 0.26 (0.29) | 0.29 (0.22) | 0.48 (0.58) | 0.36 (0.30) | 0.16 (0.11) | 0.19 (0.10) |
  Cycle 1 Day 15 (336 hours Post-dose): number analyzed (Participants) | 5 | 2 | 4 | 4 | 4 | 5 | 3 | 0
  Cycle 1 Day 15 (336 hours Post-dose) | 1.20 (0.92) | 0.97 (0.16) | 0.42 (0.38) | 4.24 (7.89) | 0.39 (0.29) | 0.33 (0.29) | 0.27 (0.19) |

ADVERSE EVENTS:
Time Frame: Part 1: AEs: From Day 1 up to the end of safety follow-up (up to 28.5 months) All-cause Mortality: Part 1: From Day 1 up to end of survival follow-up (36 months) Part 2: AEs and All-cause Mortality: From Day 1 up to the end of safety follow-up (up to 9.3 months)
Description: Safety population included all participants who received at least one dose of study treatment, whether prematurely withdrawn from the study or not.
Arm/Group | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg
All-Cause Mortality (participants affected / at risk) | 5/6 | 4/6 | 4/7 | 5/7 | 5/7 | 3/6 | 3/7 | 2/3
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 3/7 | 2/7 | 4/7 | 1/6 | 4/7 | 1/3
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 7/7 | 7/7 | 7/7 | 5/6 | 7/7 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg (N=6) | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg (N=6) | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg (N=7) | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg (N=7) | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg (N=7) | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg (N=6) | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg (N=7) | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune system disorder (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid sinus syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Cohort 1 - RO7296682 0.3 mg + Atezolizumab 1200 mg (N=6) | Part 1: Cohort 2 - RO7296682 1.5 mg + Atezolizumab 1200 mg (N=6) | Part 1: Cohort 3 - RO7296682 9 mg + Atezolizumab 1200 mg (N=7) | Part 1: Cohort 4 - RO7296682 20 mg + Atezolizumab 1200 mg (N=7) | Part 1: Cohort 5 - RO7296682 40 mg + Atezolizumab 1200 mg (N=7) | Part 1: Cohort 6 - RO7296682 80 mg + Atezolizumab 1200 mg (N=6) | Part 1: Cohort 7 - RO7296682 160 mg + Atezolizumab 1200 mg (N=7) | Part 2: Cohort 1 - RO7296682 70 mg + Atezolizumab 1200 mg (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scleral haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breath odour (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 3 (4) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (5) | 2 (4) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 3 (4) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Oral pruritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (7) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 3 (4) | 1 (1) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (3) | 2 (2) | 5 (5) | 1 (1) | 4 (6) | 1 (1) | 0 (0)
Mucosal dryness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Necrosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (6) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Campylobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access site erythema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Secondary cerebellar degeneration (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (5) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillar ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (5) | 5 (7) | 4 (5) | 4 (4) | 3 (6) | 1 (1) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (3) | 2 (3) | 6 (8) | 2 (2) | 3 (6) | 1 (2) | 2 (3)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (5) | 1 (1) | 2 (2) | 2 (4) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT04642365/Prot_SAP_000.pdf